CLINICAL TRIAL: NCT05741294
Title: Open Phase IV Study to Assess the Impact of Tirbanibulin on the Wellbeing of Patients With Actinic Keratoses (TIRBASKIN)
Brief Title: A Study of Tirbanibulin on the Wellbeing of Participants With Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-14789-42; 2022-001251-16 (EudraCT Number)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Actinic Keratosis
Keywords: Keratosis; Tirbanibulin
MeSH Terms: conditions — Keratosis, Actinic; Keratosis | interventions — tirbanibulin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirbanibulin 2.5 milligrams (mg) ointment (Experimental): Participants will apply tirbanibulin ointment- topically at a dose of 2.5 mg once daily for 5 consecutive days- on the face or scalp.
  Interventions: Drug: Tirbanibulin 2.5 mg ointment

INTERVENTIONS:
Drug: Tirbanibulin 2.5 mg ointment — Participants will apply tirbanibulin 2.5 mg ointment topically for 5 consecutive days over 25 square centimeters (cm^2) of the face or scalp.

SUMMARY:
The purpose of the study is to assess treatment satisfaction on Day 57 in participants with Actinic Keratoses (AK) of the face or scalp following treatment with tirbanibulin ointment 1 percent (%) administered once daily for 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Males or females aged greater than or equal to (>=)18 years.
3. Diagnosis of clinically typical AK in one contiguous area on the face or scalp with a treatment area of 25^cm2 containing 4-8 AK lesions.
4. Participants not previously treated for AK on the current treatment area of the face or scalp in the last 6 months. However, previous AK treatment in other small areas (up to 25^cm2) in the last greater than >1 to less than <6 months is allowed.
5. Females must be postmenopausal (A female said to be postmenopausal should be >45 years of age with at least 12 months of amenorrhea), surgically sterile (by hysterectomy, bilateral oophorectomy, or tubal ligation); or, if of child-bearing potential, must be using highly effective contraception for at least 30 days or 1 menstrual cycle, whichever is longer, prior to study treatment and must agree to continue to use highly effective contraception for at least 30 days following their last dose of study treatment. Highly effective contraception includes oral hormonal contraceptives, hormonal contraceptive intercourse.
6. Sexually active males who have not had a vasectomy, and whose partner is reproductively capable, must agree to use barrier contraception from Screening through 90 days after their last dose of study treatment.
7. All participants must agree not to donate sperm or eggs from screening through 90 days following their last dose of study treatment.
8. Females of child-bearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 0 prior to dose administration.
9. Willing to avoid excessive sun or UV (ultraviolet light) light exposure to the face or scalp.

Exclusion Criteria:

1. Clinically atypical and/or rapidly changing AK lesions.
2. Location of the treatment area is within 5 cm of an incompletely healed wound or a suspected basal cell carcinoma (BCC)/squamous cell carcinoma (SCC).
3. Skin disease (e.g., atopic dermatitis, psoriasis, eczema) or condition (e.g., open wounds, scarring) in the treatment area that might interfere with the study results or suppose an unacceptable risk.
4. History of sensitivity to any of the ingredients in the tirbanibulin formulation.
5. Participated in a clinical trial during which an investigational study medication was administered within 30 days or 5 half-lives of the investigational product, whichever is longer, before dosing.
6. Participants with a history of tirbanibulin treatment for AK lesions and participants who are currently on tirbanibulin treatment for AK lesions.
7. Use of immunomodulators (e.g., azathioprine), cytotoxic drugs (e.g., cyclophosphamide, vinblastine, chlorambucil, methotrexate) or interferons/ interferon inducers and systemic immunosuppressive agents (e.g., cyclosporine, prednisone, methotrexate, alefacept, infliximab) within 4 weeks prior to the Screening visit, except for organ transplant recipients under stable immunosuppressive therapy for 6 months.
8. Use of systemic retinoids (e.g., isotretinoin, acitretin, bexarotene) within 6 months prior to the Screening visit.
9. Use of the following therapies and/or medications within 2 weeks prior to the Screening Visit:

   * Cosmetic or therapeutic procedures (e.g., use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within the treatment area or within 2 cm of the selected treatment area
   * Acid-containing therapeutic products (e.g., salicylic acid or fruit acids, such as alpha- and beta-hydroxyl acids and glycolic acids), topical retinoids, or light chemical peels within the treatment area or within 2 cm of the selected treatment area
   * Topical salves (nonmedicated/nonirritant lotion and cream are acceptable) or topical steroids within the treatment area or within 2 cm of the selected treatment area; artificial tanners within the treatment area or within 5 cm of the selected treatment area.
10. Females who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Lecchi, Study Director — Almirall, srl
Locations (37):
- Italy (7):
  - Almirall Investigational Site 1, Cagliari
  - Almirall Investigational Site 2, Catania
  - Almirall Investigational Site 3, Napoli
  - Almirall Investigational Site 4, Pisa
  - Almirall Investigational Site 5, Rimini
  - Almirall Investigational Site 6, Torino
  - Almirall Investigational Site 7, Trieste
- Spain (30):
  - Almirall Investigational Site 1, Alcorcón
  - Almirall Investigational Site 2, Alicante
  - Almirall Investigational Site 3, Badalona
  - Almirall Investigational Site 4, Barcelona
  - Almirall Investigational Site 5, Barcelona
  - Almirall Investigational Site 6, Barcelona
  - Almirall Investigational Site 7, Barcelona
  - Almirall Investigational Site 8, Bilbao
  - Almirall Investigational Site 9, Córdoba
  - Almirall Investigational Site 10, Fuenlabrada
  - Almirall Investigational Site 11, Granada
  - Almirall Investigational Site 12, Madrid
  - Almirall Investigational Site 13, Madrid
  - Almirall Investigational Site 14, Madrid
  - Almirall Investigational Site 15, Madrid
  - Almirall Investigational Site 16, Majadahonda
  - Almirall Investigational Site 17, Málaga
  - Almirall Investigational Site 18, Palma
  - Almirall Investigational Site 19, Pontevedra
  - Almirall Investigational Site 20, Sabadell
  - Almirall Investigational Site 21, Salamanca
  - Almirall Investigational Site 22, Santa Cruz de Tenerife
  - Almirall Investigational Site 23, Seville
  - Almirall Investigational Site 24, Seville
  - Almirall Investigational Site 25, Valencia
  - Almirall Investigational Site 26, Valencia
  - Almirall Investigational Site 27, Valencia
  - Almirall Investigational Site 28, Vigo
  - Almirall Investigational Site 29, Zaragoza
  - Almirall Investigational Site 30, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 37 sites in Europe (7 in Italy and 30 in Spain) from 20 January 2023 to 19 January 2024.
Pre-assignment Details: A total of 340 participants were screened, of which 334 participants enrolled in this study.
Groups:
- Tirbanibulin 2.5 mg: Participants applied tirbanibulin ointment- topically at a dose of 2.5 milligrams (mg) once daily for 5 consecutive days on the face or scalp.
Period: Overall Study
Arm/Group | Tirbanibulin 2.5 mg
Started | 334
Evaluable Population (Evaluable population consisted of FAS participants who completed the 57 days of observation and have the TSQM-9 assessment) | 328
Line-field Confocal Optical Coherence Tomography (LC-OCT) Population (LC-OCT population consisted of FAS participants who performed at least one valid LC-OCT assessment.) | 12
Safety Population (Safety population consisted of FAS participants.) | 334
Completed | 327
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Protocol deviation | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all participants who signed the informed consent form and applied at least one dose of tirbanibulin.
Groups:
- Tirbanibulin 2.5 mg: Participants applied tirbanibulin ointment- topically at a dose of 2.5 mg once daily for 5 consecutive days on the face or scalp.
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 278
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 334

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Questionnaire for Medication Version 9 (TSQM-9) Total Score of Each Components at Day 57
Description: TSQM-9 was a 9-item clinically validated psychometric instrument developed from the TSQM 1.4. TSQM-9 measures participant satisfaction with the medication in 3 domains: Effectiveness, convenience, and global satisfaction. The scores were computed by adding items for each domain, i.e., 1 to 3 for effectiveness, 4 to 6 for convenience, and 7 to 9 for global satisfaction. The lowest possible score (1 for each item and 3 for all 3 subscales) was subtracted from the composite score and divided by the greatest possible score range. The greatest range was (7-1) x 3 items = 18 for effectiveness and convenience, and (5-1) x 3 items = 12 for global satisfaction. This provided a transformed score between 0 and 1 that was then multiplied by 100. TSQM-9 domain scores range from 0 to 100, with higher scores indicating greater satisfaction for that domain. A positive change from baseline indicates improvement.
Time Frame: At Day 57
Population: Evaluable population consisted of FAS participants who completed the 57 days of observation and have the TSQM-9 assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
score on a scale
  Effectiveness Total Score Value | 73.64 [71.28 to 76.01]
  Convenience Total Score Value | 82.81 [81.28 to 84.34]
  Global Satisfaction Total Score Value | 76.94 [74.89 to 78.99]

2. Secondary Outcome: Change From Baseline in Skindex-16 Questionnaire Symptoms Sub-Score at Day 57
Description: Skindex-16 was used for participants to rate skin conditions that have occurred within the previous week. The Skindex-16 consisted of 16 items that were divided into three sub-scores: Symptoms (four items, range 0-24), Emotions (seven items, range 0-42), and Functioning (five items, range 0-30). Participant were asked to respond on how much their skin condition bothered them in the week prior to administration of the Skindex-16. Each item was scored on a scale ranged from 0 (never bothered) to 6 (always bothered), where higher score indicated continued/more botheration. Item scores are transformed to 0 to 100 scale, and domain scores are calculated as the average of the item scores comprising the domain. Net positive changes in respective subscale scoring indicates improvement in that particular quality of life assessment (i.e., Symptoms, Emotions, Functioning), while net negative changes in scoring indicates decrease in that particular quality of life assessment.
Time Frame: Baseline, Day 57
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
score on a scale
  Symptoms Sub-Score: Change at Day 57 | -10.49 [-12.55 to -8.44]
  Emotions Sub-Score: Change at Day 57 | -11.56 [-13.56 to -9.55]
  Functioning Sub-Score: Change at Day 57 | -2.49 [-3.98 to -1.00]

3. Secondary Outcome: Percentage of Participants With Organoleptic Properties of Tirbanibulin Assessed on a Likert Scale at Day 8
Description: Likert scale was an instrument used to measure the individual's degree of agreement and disagreement with a variety of statements about some attitude, options, or their feelings. In this study, the product's organoleptic properties are evaluated with Likert scale. The questionnaire was built with questions related to the product's characteristics namely appearance, color, convenience, texture, smell, and the feelings experienced during drug application. The Likert scale offers 7 possible answers, from "totally agree",' In agreement", "Somewhat agree", "Neither agree nor disagree", "Something in disagreement", "In disagreement" and "totally in disagreement".
Time Frame: At Day 8
Population: Evaluable population consisted of FAS participants who completed the 57 days of observation and have the TSQM-9 assessment. Here, "Overall number of Participants" signifies participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 327
Percentage of participants
  The general appearance of the product is good: Totally agree | 52.60 [43.75 to 61.34]
  The general appearance of the product is good: In agreement | 38.23 [29.91 to 47.04]
  The general appearance of the product is good: Somewhat agree | 3.06 [0.85 to 7.22]
  The general appearance of the product is good: Neither agree nor disagree | 5.20 [2.11 to 10.15]
  The general appearance of the product is good: Something in disagreement | 0.31 [0.00 to 2.76]
  The general appearance of the product is good: In disagreement | 0.61 [0.00 to 3.36]
  The general appearance of the product is good: Totally in disagreement | 0 [0 to 0]
  The overall assessment of the product is very satisfactory: Totally agree | 36.70 [27.64 to 46.33]
  The overall assessment of the product is very satisfactory: In agreement | 38.53 [29.35 to 48.21]
  The overall assessment of the product is very satisfactory: Somewhat agree | 8.26 [3.75 to 14.57]
  The overall assessment of the product is very satisfactory: Neither agree nor disagree | 10.40 [5.28 to 17.23]
  The overall assessment of the product is very satisfactory: Something in disagreement | 1.53 [0.00 to 5.18]
  The overall assessment of the product is very satisfactory: In disagreement | 3.36 [0.74 to 8.01]
  The overall assessment of the product is very satisfactory: Totally in disagreement | 1.22 [0.00 to 4.66]
  I would recommend the product: Totally agree | 34.86 [25.95 to 44.43]
  I would recommend the product: In agreement | 33.64 [24.83 to 43.15]
  I would recommend the product: Somewhat agree | 5.81 [2.13 to 11.40]
  I would recommend the product: Neither agree nor disagree | 18.04 [11.25 to 26.22]
  I would recommend the product: Something in disagreement | 1.22 [0.00 to 4.66]
  I would recommend the product: In disagreement | 3.06 [0.59 to 7.56]
  I would recommend the product: Totally in disagreement | 3.36 [0.74 to 8.01]
  The color of the product is nice: Totally agree | 36.70 [29.37 to 44.55]
  The color of the product is nice: In agreement | 36.09 [28.80 to 43.92]
  The color of the product is nice: Somewhat agree | 5.81 [2.90 to 10.47]
  The color of the product is nice: Neither agree nor disagree | 20.80 [14.96 to 27.79]
  The color of the product is nice: Something in disagreement | 0 [0 to 0]
  The color of the product is nice: In disagreement | 0.61 [0.02 to 3.17]
  The color of the product is nice: Totally in disagreement | 0 [0 to 0]
  The texture of the product is nice: Totally agree | 48.93 [40.14 to 57.76]
  The texture of the product is nice: In agreement | 40.37 [31.92 to 49.21]
  The texture of the product is nice: Somewhat agree | 5.20 [2.11 to 10.15]
  The texture of the product is nice: Neither agree nor disagree | 4.28 [1.54 to 8.93]
  The texture of the product is nice: Something in disagreement | 0.61 [0.00 to 3.36]
  The texture of the product is nice: In disagreement | 0.61 [0.00 to 3.36]
  The texture of the product is nice: Totally in disagreement | 0 [0 to 0]
  The texture of the product is watery: Totally agree | 12.84 [7.12 to 20.18]
  The texture of the product is watery: In agreement | 18.65 [11.76 to 26.91]
  The texture of the product is watery: Somewhat agree | 9.79 [4.83 to 16.48]
  The texture of the product is watery: Neither agree nor disagree | 15.90 [9.52 to 23.76]
  The texture of the product is watery: Something in disagreement | 8.26 [3.75 to 14.57]
  The texture of the product is watery: In disagreement | 19.88 [12.77 to 28.29]
  The texture of the product is watery: Totally in disagreement | 14.68 [8.54 to 22.34]
  The texture of the product is oily: Totally agree | 11.31 [5.96 to 18.35]
  The texture of the product is oily: In agreement | 15.90 [9.52 to 23.76]
  The texture of the product is oily: Somewhat agree | 9.48 [4.61 to 16.10]
  The texture of the product is oily: Neither agree nor disagree | 16.82 [10.26 to 24.82]
  The texture of the product is oily: Something in disagreement | 6.73 [2.72 to 12.61]
  The texture of the product is oily: In disagreement | 20.49 [13.28 to 28.97]
  The texture of the product is oily: Totally in disagreement | 19.27 [12.26 to 27.60]
  The texture of the product is creamy: Totally agree | 40.06 [30.78 to 49.77]
  The texture of the product is creamy: In agreement | 41.28 [31.93 to 51.01]
  The texture of the product is creamy: Somewhat agree | 7.03 [2.92 to 13.00]
  The texture of the product is creamy: Neither agree nor disagree | 7.34 [3.13 to 13.40]
  The texture of the product is creamy: Something in disagreement | 1.53 [0.00 to 5.18]
  The texture of the product is creamy: In disagreement | 1.83 [0.08 to 5.68]
  The texture of the product is creamy: Totally in disagreement | 0.92 [0.00 to 4.11]
  The skin was greasy after applying the treatment: Totally agree | 12.84 [7.12 to 20.18]
  The skin was greasy after applying the treatment: In agreement | 25.08 [17.20 to 34.03]
  The skin was greasy after applying the treatment: Somewhat agree | 14.68 [8.54 to 22.34]
  The skin was greasy after applying the treatment: Neither agree nor disagree | 8.56 [3.96 to 14.95]
  The skin was greasy after applying the treatment: Something in disagreement | 3.98 [1.06 to 8.89]
  The skin was greasy after applying the treatment: In disagreement | 17.13 [10.50 to 25.17]
  The skin was greasy after applying the treatment: Totally in disagreement | 17.74 [11.00 to 25.87]
  The smell of the product is pleasant: Totally agree | 23.85 [16.14 to 32.70]
  The smell of the product is pleasant: In agreement | 23.55 [15.88 to 32.36]
  The smell of the product is pleasant: Somewhat agree | 7.65 [3.33 to 13.79]
  The smell of the product is pleasant: Neither agree nor disagree | 42.51 [33.09 to 52.25]
  The smell of the product is pleasant: Something in disagreement | 0.61 [0.00 to 3.53]
  The smell of the product is pleasant: In disagreement | 0.92 [0.00 to 4.11]
  The smell of the product is pleasant: Totally in disagreement | 0.92 [0.00 to 4.11]
  The product feels pleasant on the skin: Totally agree | 27.22 [19.07 to 36.35]
  The product feels pleasant on the skin: In agreement | 30.28 [21.79 to 39.61]
  The product feels pleasant on the skin: Somewhat agree | 10.70 [5.50 to 17.60]
  The product feels pleasant on the skin: Neither agree nor disagree | 21.10 [13.80 to 29.66]
  The product feels pleasant on the skin: Something in disagreement | 1.83 [0.08 to 5.68]
  The product feels pleasant on the skin: In disagreement | 5.50 [1.95 to 10.99]
  The product feels pleasant on the skin: Totally in disagreement | 3.36 [0.74 to 8.01]
  The feel of the product on the skin is refreshing: Totally agree | 18.35 [11.50 to 26.56]
  The feel of the product on the skin is refreshing: In agreement | 20.80 [13.54 to 29.32]
  The feel of the product on the skin is refreshing: Somewhat agree | 11.31 [5.96 to 18.35]
  The feel of the product on the skin is refreshing: Neither agree nor disagree | 22.94 [15.36 to 31.69]
  The feel of the product on the skin is refreshing: Something in disagreement | 5.81 [2.13 to 11.40]
  The feel of the product on the skin is refreshing: In disagreement | 10.09 [5.06 to 16.86]
  The feel of the product on the skin is refreshing: Totally in disagreement | 10.70 [5.50 to 17.60]
  The product offers a protective feeling: Totally agree | 20.80 [13.54 to 29.32]
  The product offers a protective feeling: In agreement | 25.38 [17.47 to 34.36]
  The product offers a protective feeling: Somewhat agree | 9.48 [4.61 to 16.10]
  The product offers a protective feeling: Neither agree nor disagree | 30.28 [21.79 to 39.61]
  The product offers a protective feeling: Something in disagreement | 3.06 [0.59 to 7.56]
  The product offers a protective feeling: In disagreement | 5.81 [2.13 to 11.40]
  The product offers a protective feeling: Totally in disagreement | 5.20 [1.76 to 10.58]
  The product is easy to apply: Totally agree | 66.36 [56.85 to 75.17]
  The product is easy to apply: In agreement | 27.22 [19.07 to 36.35]
  The product is easy to apply: Somewhat agree | 3.67 [0.89 to 8.45]
  The product is easy to apply: Neither agree nor disagree | 0.92 [0.00 to 4.11]
  The product is easy to apply: Something in disagreement | 0.92 [0.00 to 4.11]
  The product is easy to apply: In disagreement | 0.31 [0.00 to 2.90]
  The product is easy to apply: Totally in disagreement | 0.61 [0.00 to 3.53]
  The product can be distributed evenly and easily: Totally agree | 64.53 [55.79 to 72.66]
  The product can be distributed evenly and easily: In agreement | 29.05 [21.48 to 37.50]
  The product can be distributed evenly and easily: Somewhat agree | 4.28 [1.54 to 8.93]
  The product can be distributed evenly and easily: Neither agree nor disagree | 0.61 [0.00 to 3.36]
  The product can be distributed evenly and easily: Something in disagreement | 0.92 [0.00 to 3.91]
  The product can be distributed evenly and easily: In disagreement | 0.61 [0.00 to 3.36]
  The product can be distributed evenly and easily: Totally in disagreement | 0 [0 to 0]
  Product remains on application area, without spreading to neighboring areas: Totally agree | 57.19 [47.44 to 66.62]
  Product remains on application area, without spreading to neighboring areas: In agreement | 29.97 [21.52 to 39.29]
  Product remains on application area, without spreading to neighboring areas: Somewhat agree | 6.12 [2.33 to 11.81]
  Product remains on application area, without spreading to neighboring areas: Neither agree/ disagree | 2.75 [0.44 to 7.11]
  Product remains on application area without spreading to neighboring areas:Something in disagreement | 2.14 [0.19 to 6.17]
  Product remains on application area, without spreading to neighboring areas: In disagreement | 0.61 [0.00 to 3.53]
  Product remains on application area, without spreading to neighboring areas: Totally in disagreement | 1.22 [0.00 to 4.66]
  The product packaging is practical: Totally agree | 50.76 [41.06 to 60.43]
  The product packaging is practical: In agreement | 33.94 [25.11 to 43.47]
  The product packaging is practical: Somewhat agree | 6.12 [2.33 to 11.81]
  The product packaging is practical: Neither agree nor disagree | 3.06 [0.59 to 7.56]
  The product packaging is practical: Something in disagreement | 2.14 [0.19 to 6.17]
  The product packaging is practical: In disagreement | 3.36 [0.74 to 8.01]
  The product packaging is practical: Totally in disagreement | 0.61 [0.00 to 3.53]

4. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Version 1.4 (TSQM 1.4) Components Scores at Day 57
Description: TSQM 1.4 was a 14-item robust instrument that psychometrically evaluates the treatment satisfaction of the administered medication. The instrument is designed with 4 scales consisting of 14 questions. These 14 questions were derived from an original set of 55 questions extracted from exhaustive literature review and treatment groups through multistep iterative process. The 4 scales focused on effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions:12-14). Global Satisfaction- Question 12 scored as 1 (not at all confident) to 5 (extremely confident); question 13 scored as 1 (not at all certain) to 5 (extremely certain); and question 14 scored as 1 (extremely dissatisfied) to 7 (extremely satisfied). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction.
Time Frame: At Day 57
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
score on a scale
  Effectiveness score value at Day 57 | 73.64 [71.28 to 76.01]
  Convenience score value at Day 57 | 82.81 [81.28 to 84.34]
  Side Effects score value at Day 57 | 97.47 [96.59 to 98.34]
  Global satisfaction score value at Day 57 | 76.94 [74.89 to 78.99]

5. Secondary Outcome: Percentage of Patients Who Answered Expert Panel Questionnaire (EPQ) (Question 1 to Question 9) at Day 57
Description: An expert panel on consensus developed a questionnaire directed to patients consisting of 9 simple items using a qualitative modified delphi method. Expert panel agreed to ask 9 specific items; 1: Overall appearance of the skin (much worse to much improved); 2: Treatment satisfaction of skin looks (extremely dissatisfied to extremely satisfied); 3: Treatment satisfaction of skin texture (extremely dissatisfied to extremely satisfied); 4: Duration of skin reactions (much shorter to much longer); 5: rate the severity of skin reactions (much better to much worse); 6: impact on your daily activities due to skin reactions (much better to much worse); 7: rate the convenience/ease of use (much better to much worse); 8: rate your overall satisfaction (much better to much worse); 9: You need to be retreated for AK, how likely are you to consider tirbanibulin (very unlikely to very likely).
Time Frame: At Day 57
Population: Evaluable population consisted of FAS participants who completed the 57 days of observation and have the TSQM-9 assessment. Here, "number analyzed" signifies participants who were evaluable at specific category.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
Percentage of patients
  Overall appearance of the skin: Much worse: number analyzed (Participants) | 318
  Overall appearance of the skin: Much worse | 0.31 [0.00 to 2.68]
  Overall appearance of the skin: Somewhat worse: number analyzed (Participants) | 318
  Overall appearance of the skin: Somewhat worse | 0.31 [0.00 to 2.68]
  Overall appearance of the skin: No change: number analyzed (Participants) | 318
  Overall appearance of the skin: No change | 6.92 [3.66 to 11.94]
  Overall appearance of the skin: Somewhat improved: number analyzed (Participants) | 318
  Overall appearance of the skin: Somewhat improved | 24.84 [18.45 to 32.27]
  Overall appearance of the skin: Much improved: number analyzed (Participants) | 318
  Overall appearance of the skin: Much improved | 67.61 [59.78 to 74.72]
  Treatment satisfaction of skin looks: Extremely Dissatisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Extremely Dissatisfied | 0 [0 to 0]
  Treatment satisfaction of skin looks: Very Dissatisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Very Dissatisfied | 0.63 [0.00 to 3.45]
  Treatment satisfaction of skin looks: Dissatisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Dissatisfied | 2.83 [0.71 to 6.97]
  Treatment satisfaction of skin looks: Somewhat Satisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Somewhat Satisfied | 7.23 [3.43 to 12.86]
  Treatment satisfaction of skin looks: Satisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Satisfied | 25.79 [18.47 to 34.14]
  Treatment satisfaction of skin looks: Very Satisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Very Satisfied | 30.19 [22.40 to 38.82]
  Treatment satisfaction of skin looks: Extremely Satisfied: number analyzed (Participants) | 318
  Treatment satisfaction of skin looks: Extremely Satisfied | 33.33 [25.26 to 42.12]
  Treatment satisfaction of skin texture: Extremely Dissatisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Extremely Dissatisfied | 0 [0 to 0]
  Treatment satisfaction of skin texture: Very Dissatisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Very Dissatisfied | 1.25 [0.05 to 4.51]
  Treatment satisfaction of skin texture: Dissatisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Dissatisfied | 2.80 [0.70 to 6.91]
  Treatment satisfaction of skin texture: Somewhat Satisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Somewhat Satisfied | 7.17 [3.40 to 12.75]
  Treatment satisfaction of skin texture: Satisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Satisfied | 30.84 [23.03 to 39.47]
  Treatment satisfaction of skin texture: Very Satisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Very Satisfied | 27.73 [20.23 to 36.17]
  Treatment satisfaction of skin texture: Extremely Satisfied: number analyzed (Participants) | 321
  Treatment satisfaction of skin texture: Extremely Satisfied | 30.22 [22.46 to 38.81]
  Duration of skin reactions: Much shorter: number analyzed (Participants) | 186
  Duration of skin reactions: Much shorter | 44.62 [34.53 to 55.09]
  Duration of skin reactions: Somewhat shorter: number analyzed (Participants) | 186
  Duration of skin reactions: Somewhat shorter | 23.66 [15.73 to 33.40]
  Duration of skin reactions: Same: number analyzed (Participants) | 186
  Duration of skin reactions: Same | 18.82 [11.74 to 28.04]
  Duration of skin reactions: Somewhat longer: number analyzed (Participants) | 186
  Duration of skin reactions: Somewhat longer | 9.14 [4.42 to 16.67]
  Duration of skin reactions: Much longer: number analyzed (Participants) | 186
  Duration of skin reactions: Much longer | 3.76 [1.11 to 9.60]
  Rate the severity of skin reactions: Much better: number analyzed (Participants) | 187
  Rate the severity of skin reactions: Much better | 51.34 [40.98 to 61.60]
  Rate the severity of skin reactions: Somewhat better: number analyzed (Participants) | 187
  Rate the severity of skin reactions: Somewhat better | 21.93 [14.30 to 31.47]
  Rate the severity of skin reactions: Same: number analyzed (Participants) | 187
  Rate the severity of skin reactions: Same | 16.58 [9.97 to 25.48]
  Rate the severity of skin reactions: Somewhat worse: number analyzed (Participants) | 187
  Rate the severity of skin reactions: Somewhat worse | 8.02 [3.68 to 15.24]
  Rate the severity of skin reactions: Much worse: number analyzed (Participants) | 187
  Rate the severity of skin reactions: Much worse | 2.14 [0.37 to 7.18]
  Impact on your daily activities due to skin reactions: Much better: number analyzed (Participants) | 189
  Impact on your daily activities due to skin reactions: Much better | 49.74 [39.48 to 60.00]
  Impact on your daily activities due to skin reactions: Somewhat better: number analyzed (Participants) | 189
  Impact on your daily activities due to skin reactions: Somewhat better | 13.76 [7.81 to 22.16]
  Impact on your daily activities due to skin reactions: Same: number analyzed (Participants) | 189
  Impact on your daily activities due to skin reactions: Same | 31.75 [22.79 to 41.94]
  Impact on your daily activities due to skin reactions: Somewhat worse: number analyzed (Participants) | 189
  Impact on your daily activities due to skin reactions: Somewhat worse | 3.70 [1.09 to 9.46]
  Impact on your daily activities due to skin reactions: Much worse: number analyzed (Participants) | 189
  Impact on your daily activities due to skin reactions: Much worse | 1.06 [0.04 to 5.39]
  Rate the convenience/ease of use: Much better: number analyzed (Participants) | 207
  Rate the convenience/ease of use: Much better | 57.97 [48.02 to 67.42]
  Rate the convenience/ease of use: Somewhat better: number analyzed (Participants) | 207
  Rate the convenience/ease of use: Somewhat better | 19.81 [12.86 to 28.63]
  Rate the convenience/ease of use: Same: number analyzed (Participants) | 207
  Rate the convenience/ease of use: Same | 19.81 [12.86 to 28.63]
  Rate the convenience/ease of use: Somewhat worse: number analyzed (Participants) | 207
  Rate the convenience/ease of use: Somewhat worse | 1.93 [0.34 to 6.51]
  Rate the convenience/ease of use: Much worse: number analyzed (Participants) | 207
  Rate the convenience/ease of use: Much worse | 0.48 [0.00 to 4.08]
  Rate your overall satisfaction: Much better: number analyzed (Participants) | 209
  Rate your overall satisfaction: Much better | 60.29 [50.40 to 69.54]
  Rate your overall satisfaction: Somewhat better: number analyzed (Participants) | 209
  Rate your overall satisfaction: Somewhat better | 21.53 [14.32 to 30.49]
  Rate your overall satisfaction: Same: number analyzed (Participants) | 209
  Rate your overall satisfaction: Same | 13.40 [7.77 to 21.28]
  Rate your overall satisfaction: Somewhat worse: number analyzed (Participants) | 209
  Rate your overall satisfaction: Somewhat worse | 3.83 [1.24 to 9.26]
  Rate your overall satisfaction: Much worse: number analyzed (Participants) | 209
  Rate your overall satisfaction: Much worse | 0.96 [0.04 to 4.89]
  You need to be retreated for AK, how likely to consider tirbanibulin: Very unlikely | 3.66 [1.49 to 7.67]
  You need to be retreated for AK, how likely to consider tirbanibulin: Somewhat unlikely | 2.44 [0.78 to 5.98]
  You need to be retreated for AK, how likely to consider tirbanibulin: Neutral | 7.62 [4.21 to 12.72]
  You need to be retreated for AK, how likely to consider tirbanibulin: Somewhat likely | 18.60 [13.08 to 25.37]
  You need to be retreated for AK, how likely to consider tirbanibulin: Very likely | 67.68 [59.98 to 74.69]

6. Secondary Outcome: Percentage of Physician Who Answered Expert Panel Questionnaire (EPQ) (Question 1 to Question 10) at Day 57
Description: An expert panel on consensus developed a questionnaire directed to physicians consisting of 10 simple items using a qualitative modified delphi method. Expert panel agreed to ask 10 specific items-1: Overall appearance of the skin (much worse to much improved); 2: Treatment satisfaction of skin looks (extremely dissatisfied to extremely satisfied); 3: Treatment satisfaction of skin texture (extremely dissatisfied to extremely satisfied); 4: Duration of skin reactions (much shorter to much longer); 5: rate the severity of skin reactions (much better to much worse); 6: impact on patient's daily activities due to skin reactions (much better to much worse); 7: rate the convenience/ease of use (much better to much worse); 8: rate your overall satisfaction (much better to much worse); 9: patient needs to be retreated for AK, how likely to consider tirbanibulin (very unlikely to very likely);10: severity of skin photodamage in the original AK treated area (absent to severe).
Time Frame: At Day 57
Population: Evaluable population consisted of FAS participants who completed the 57 days of observation and have the TSQM-9 assessment. Here, "Overall number of Participants" signifies participants who were evaluable for this outcome and "number analyzed" signifies participants who were evaluable at specific category.
Measure: Number (95% Confidence Interval); unit: Percentage of physician
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 326
Percentage of physician
  Overall appearance of the skin:Much worse | 1.23 [0.21 to 4.19]
  Overall appearance of the skin: Somewhat worse | 1.23 [0.21 to 4.19]
  Overall appearance of the skin: No change | 1.23 [0.21 to 4.19]
  Overall appearance of the skin: Somewhat improved | 21.78 [15.81 to 28.87]
  Overall appearance of the skin: Much improved | 74.54 [67.17 to 80.93]
  Treatment satisfaction of skin looks: Extremely Dissatisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Extremely Dissatisfied | 0.31 [0.00 to 2.93]
  Treatment satisfaction of skin looks: Very Dissatisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Very Dissatisfied | 0.31 [0.00 to 2.93]
  Treatment satisfaction of skin looks: Dissatisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Dissatisfied | 0.31 [0.00 to 2.93]
  Treatment satisfaction of skin looks: Somewhat Satisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Somewhat Satisfied | 6.79 [2.75 to 12.72]
  Treatment satisfaction of skin looks: Satisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Satisfied | 25.31 [17.37 to 34.33]
  Treatment satisfaction of skin looks: Very Satisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Very Satisfied | 31.48 [22.84 to 40.93]
  Treatment satisfaction of skin looks: Extremely Satisfied: number analyzed (Participants) | 324
  Treatment satisfaction of skin looks: Extremely Satisfied | 35.49 [26.49 to 45.13]
  Treatment satisfaction of skin texture: Extremely Dissatisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Extremely Dissatisfied | 0.31 [0.00 to 2.92]
  Treatment satisfaction of skin texture: Very Dissatisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Very Dissatisfied | 0.31 [0.00 to 2.92]
  Treatment satisfaction of skin texture: Dissatisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Dissatisfied | 0.92 [0.00 to 4.14]
  Treatment satisfaction of skin texture: Somewhat Satisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Somewhat Satisfied | 6.77 [2.74 to 12.68]
  Treatment satisfaction of skin texture: Satisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Satisfied | 27.69 [19.47 to 36.89]
  Treatment satisfaction of skin texture: Very Satisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Very Satisfied | 32.92 [24.16 to 42.43]
  Treatment satisfaction of skin texture: Extremely Satisfied: number analyzed (Participants) | 325
  Treatment satisfaction of skin texture: Extremely Satisfied | 31.08 [22.49 to 40.49]
  Duration of skin reactions: Much shorter: number analyzed (Participants) | 223
  Duration of skin reactions: Much shorter | 60.09 [50.51 to 69.08]
  Duration of skin reactions: Somewhat shorter: number analyzed (Participants) | 223
  Duration of skin reactions: Somewhat shorter | 27.35 [19.54 to 36.48]
  Duration of skin reactions: Same: number analyzed (Participants) | 223
  Duration of skin reactions: Same | 8.52 [4.29 to 15.14]
  Duration of skin reactions: Somewhat longer: number analyzed (Participants) | 223
  Duration of skin reactions: Somewhat longer | 3.14 [0.92 to 8.06]
  Duration of skin reactions: Much longer: number analyzed (Participants) | 223
  Duration of skin reactions: Much longer | 0.90 [0.03 to 4.60]
  Rate the severity of skin reactions: Much better: number analyzed (Participants) | 222
  Rate the severity of skin reactions: Much better | 64.86 [55.36 to 73.15]
  Rate the severity of skin reactions: Somewhat better: number analyzed (Participants) | 222
  Rate the severity of skin reactions: Somewhat better | 22.07 [14.96 to 30.80]
  Rate the severity of skin reactions: Same: number analyzed (Participants) | 222
  Rate the severity of skin reactions: Same | 9.01 [4.63 to 15.76]
  Rate the severity of skin reactions: Somewhat worse: number analyzed (Participants) | 222
  Rate the severity of skin reactions: Somewhat worse | 3.60 [1.16 to 8.74]
  Rate the severity of skin reactions: Much worse: number analyzed (Participants) | 222
  Rate the severity of skin reactions: Much worse | 0.45 [0.00 to 3.81]
  Impact on patient's daily activities due to skin reactions: Much better: number analyzed (Participants) | 214
  Impact on patient's daily activities due to skin reactions: Much better | 59.81 [50.04 to 69.00]
  Impact on patient's daily activities due to skin reactions: Somewhat better: number analyzed (Participants) | 214
  Impact on patient's daily activities due to skin reactions: Somewhat better | 19.63 [12.81 to 28.27]
  Impact on patient's daily activities due to skin reactions: Same: number analyzed (Participants) | 214
  Impact on patient's daily activities due to skin reactions: Same | 19.63 [12.81 to 28.27]
  Impact on patient's daily activities due to skin reactions: Somewhat worse: number analyzed (Participants) | 214
  Impact on patient's daily activities due to skin reactions: Somewhat worse | 0.47 [0.00 to 3.95]
  Impact on patient's daily activities due to skin reactions: Much worse: number analyzed (Participants) | 214
  Impact on patient's daily activities due to skin reactions: Much worse | 0.47 [0.00 to 3.95]
  Rate the convenience/ease of use: Much better: number analyzed (Participants) | 225
  Rate the convenience/ease of use: Much better | 65.78 [57.55 to 73.16]
  Rate the convenience/ease of use: Somewhat better: number analyzed (Participants) | 225
  Rate the convenience/ease of use: Somewhat better | 25.33 [18.82 to 33.17]
  Rate the convenience/ease of use: Same: number analyzed (Participants) | 225
  Rate the convenience/ease of use: Same | 5.33 [2.66 to 10.42]
  Rate the convenience/ease of use: Somewhat worse: number analyzed (Participants) | 225
  Rate the convenience/ease of use: Somewhat worse | 3.56 [1.52 to 8.10]
  Rate the convenience/ease of use: Much worse: number analyzed (Participants) | 225
  Rate the convenience/ease of use: Much worse | 0 [0 to 0]
  Rate your overall satisfaction: Much better: number analyzed (Participants) | 227
  Rate your overall satisfaction: Much better | 50.66 [41.25 to 60.03]
  Rate your overall satisfaction: Somewhat better: number analyzed (Participants) | 227
  Rate your overall satisfaction: Somewhat better | 37.00 [28.30 to 46.45]
  Rate your overall satisfaction: Same: number analyzed (Participants) | 227
  Rate your overall satisfaction: Same | 11.01 [6.14 to 18.11]
  Rate your overall satisfaction: Somewhat worse: number analyzed (Participants) | 227
  Rate your overall satisfaction: Somewhat worse | 0.88 [0.03 to 4.52]
  Rate your overall satisfaction: Much worse: number analyzed (Participants) | 227
  Rate your overall satisfaction: Much worse | 0.44 [0.00 to 3.73]
  Patient needs to be retreated for AK, how likely to consider tirbanibulin: Very unlikely | 3.68 [1.50 to 7.71]
  Patient needs to be retreated for AK, how likely to consider tirbanibulin: Somewhat unlikely | 1.53 [0.34 to 4.66]
  Patient needs to be retreated for AK, how likely to consider tirbanibulin: Neutral | 7.67 [4.24 to 12.79]
  Patient needs to be retreated for AK, how likely to consider tirbanibulin: Somewhat likely | 23.01 [16.89 to 30.20]
  Patient needs to be retreated for AK, how likely to consider tirbanibulin: Very likely | 64.11 [56.26 to 71.39]
  Severity of skin photodamage in the original AK treated area: Absent | 24.85 [19.38 to 31.26]
  Severity of skin photodamage in the original AK treated area: Mild | 46.63 [39.85 to 53.53]
  Severity of skin photodamage in the original AK treated area: Moderate | 27.61 [21.89 to 34.17]
  Severity of skin photodamage in the original AK treated area: Severe | 0.92 [0.24 to 3.44]

7. Secondary Outcome: Percentage of Participants With Complete (100%) Clearance of All Lesions Within the Application Area at Day 57
Description: Complete clearance of all AK lesions within the application area, is defined as a reduction from baseline in the number of lesions = 100% at Day 57. Percentage of participants with complete clearance with a reduction of 100% (i.e., clearance percentage = 100% from Baseline) in the number of lesions within the application area were reported.
Time Frame: At Day 57
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
Percentage of participants | 54.27 [48.71 to 59.75]

8. Secondary Outcome: Percentage of Participants With Partial Clearance (Reduction of at Least >=75% to <100%) of All Lesions Within the Application Area at Day 57
Description: Participants with partial clearance were patients with a reduction of >=75% (i.e., clearance percentage <=-75% from Baseline) to <100% in the number of lesions within the application area at final visit.
Time Frame: At Day 57
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
Percentage of participants | 22.56 [18.15 to 27.47]

9. Secondary Outcome: Percent Change From Baseline in Mean Number of Old and New AK Lesions at Day 57
Description: Percent change from baseline in number of old and new AK lesions at Day 57 was reported. Number of lesions at Day 57 was calculated considering both old and new lesions, as: N lesions at Baseline - N lesions at Day 57/ N lesions at Baseline * 100%.
Time Frame: At Day 57
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
Percent change | -82.22 (26.367)

10. Secondary Outcome: Percentage of Participants by Olsen Characterization at Baseline and Day 57
Description: The lesions in the identified treatment area will be classified based on Olsen characterization. Classification of AK lesions according to Olsen grade of baseline lesions: Olsen Grade I: Early AK appear as single or few, differently sized, rough, blurred, less visible than palpable, red, rough spots or very flat, non-edged plaques which reach into the reddish color; Olsen grade II: describes advanced AK as clearly visible and palpable, flat, and irregularly raised, with sharp or blurred boundaries, red, rough keratinized surface. If the surface is more strongly keratinized, the AK can also be white, yellow, or light brown. After scratching effects, a black or blue-black shade may appear; Olsen grade III: denotes "late" AK that have existed for a longer period of time and are firmly anchored on the lower surface, with an irregular, humpy surface, also wart-like and of different colors (white, brown, black).
Time Frame: Baseline (Day 0) and Day 57
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 328
Percentage of participants
  Olsen Grade I: Baseline | 62.80 [54.95 to 70.15]
  Olsen Grade I: Day 57 | 39.33 [30.95 to 48.15]
  Olsen Grade II: Baseline | 8.84 [5.12 to 14.19]
  Olsen Grade II: Day 57 | 3.66 [1.18 to 8.06]
  Olsen Grade III: Baseline | 0.0 [0.00 to 0.00]
  Olsen Grade III: Day 57 | 0.30 [0.00 to 2.75]

11. Secondary Outcome: Percentage of Participants Who Performed Line-field Confocal Optical Coherence Tomography (LC-OCT) for Clinical and Sub Clinical Lesions Assessment at Each Timepoint
Description: LC-OCT was a novel non-invasive imaging technique that enables in vivo visualization of the skin. It has been used for diagnosing and monitoring the treatment of skin disorders, including actinic keratosis. The use of LC-OCT in AK treatment progression allows for lesion classification based on histological features without the need for a biopsy. The histopathology of the skin was evaluated based on the estimated atypia score at cellular level of the LC-OCT images of clinical and subclinical lesions. Percentage of participants who performed LC-OCT for clinical and subclinical lesions assessment at each timepoint were reported.
Time Frame: Baseline, Day 8, Day 15, Day 29, and Day 57
Population: LC-OCT population consisted of FAS participants who performed at least one valid LC-OCT assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 12
Percentage of participants
  At Baseline | 100.00
  At Day 8 | 91.67
  At Day 15 | 91.67
  At Day 29 | 91.67
  At Day 57 | 100.00

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Severity of TEAEs
Description: An adverse event (AE) is as any untoward medical occurrence associated with the use of an intervention in humans after providing written informed consent for participation in the study until the end of study visit, whether considered intervention-related or not. A TEAE is defined as an AE with an onset that occurs after receiving study drug. Severity of TEAEs is graded as follows: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: From start of study administration up to Day 57
Population: Safety population consisted of FAS participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tirbanibulin 2.5 mg
Number analyzed (Participants) | 334
Participants
  Participants with TEAEs | 153
  Severity of TEAEs: Grade 1 | 132
  Severity of TEAEs: Grade 2 | 17
  Severity of TEAEs: Grade 3 | 3
  Severity of TEAEs: Grade 4 | 1

ADVERSE EVENTS:
Time Frame: From start of study administration up to Day 57
Arm/Group | Tirbanibulin 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/334
Serious Adverse Events (participants affected / at risk) | 0/334
Other Adverse Events (participants affected / at risk) | 153/334
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirbanibulin 2.5 mg (N=334)
Deafness neurosensory (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Application site hypersensitivity (General disorders) | 2
Application site pain (General disorders) | 3
Asthenia (General disorders) | 1
Burning sensation (General disorders) | 17
Chills (General disorders) | 1
Fatigue (General disorders) | 6
Inflammation (General disorders) | 1
Pain (General disorders) | 31
Temperature intolerance (General disorders) | 1
Tenderness (General disorders) | 1
Hypersensitivity (Immune system disorders) | 6
COVID 19 (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Skin injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Gout (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 13
Paraesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 5
Cellulite (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Paraesthesia (Skin and subcutaneous tissue disorders) | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 92
Skin burning sensation (Skin and subcutaneous tissue disorders) | 2
Thermal burn (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT05741294/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT05741294/SAP_001.pdf